CLINICAL TRIAL: NCT04503213
Title: Longitudinal Assessment of CSF1R-Related Leukoencephalopathy Following Stem Cell Transplantation
Brief Title: A Study to Assess CSF1R-related Leukoencephalopathy After Stem Cell Transplantation
Status: Enrolling by invitation | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Zbigniew K. Wszolek, Principal Investigator, Mayo Clinic
Other Study IDs: 20-006124
Record Dates: First submitted 2020-08-04; First posted 2020-08-07 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: CSF1R-related Leukoencephalopathy; ALSP; POLD; Hematopoietic Stem Cell Transplantation
Keywords: HDLS, Leukoencephalopathy
MeSH Terms: conditions — Hereditary Diffuse Leukoencephalopathy with Spheroids; Leukoencephalopathies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to measure the effect of Hematopoietic Stem Cell Transplantation (HSCT) on symptoms of CSF1R-related Leukoencephalopathy.

DETAILED DESCRIPTION:
The purpose of this study is to measure the effect of Hematopoietic Stem Cell Transplantation (HSCT) on symptoms of CSF1R-related Leukoencephalopathy.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age.
* Genetic confirmation of a mutation in the CSF1R gene.
* Diagnosis of CSF1R-related leukoencephalopathy.
* Anticipated to undergo haematopoietic stem cell transplantation (HSCT).

Exclusion Criteria:

* Concurrent diagnoses that may confound neuropsychological testing; e.g., major hearing/visual impairment.
* Concurrent diagnoses that may confound ambulatory measurements; e.g., amputee.
* Inability to undergo magnetic resonance imaging (MRI); e.g., MR-incompatible implant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be identified through the Mayo Clinic Florida Neurology and/or Hematology Departments. Qualifying individuals will be identified on the basis of a genetically-confirmed diagnosis of CSF1R-related leukoencephalopathy and a tentative treatment plan including haematopoietic stem cell transplantation (HSCT).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-07-21 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Improvement in cognitive and motor function | Through study completion, approximately 5 years
  Number of participants to demonstrate stability/improvements in cognitive and motor function by detailed clinical assessment and radiographic markers of disease.

CONTACTS AND LOCATIONS:
Overall Officials: Zbigniew K Wszolek, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials